CLINICAL TRIAL: NCT02774135
Title: A Prospective Cohort Study to Examine the Improvement in Preschoolers' Participation as a Result of Occupational Therapy Intervention
Brief Title: Improvement in Preschoolers' Participation as a Result of Occupational Therapy Intervention
Status: Completed | Type: Observational
Sponsor: Clalit Health Services (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Dr. Gary Leonard Robinson, Dr, MD, Pediatrics, Clalit Health Services
Other Study IDs: COM150203CTIL
Record Dates: First submitted 2016-05-09; First posted 2016-05-17 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Limited Participation in Daily Life Activities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- direct occupational therapy intervention: group will be evaluated 4 times: on referral to waiting list for treatment, before and after 9-12 direct individual treatments of 45 minutes, and follow-up after 3 months.
  Interventions: Other: direct occupational therapy intervention

INTERVENTIONS:
Other: direct occupational therapy intervention — Short term direct individual occupational therapy (9-12 weeks).Participants will receive occupational therapy intervention according to health law. The study will document the therapeutic intervention implemented in practice using the Documentation of Occupational Therapy Session during Intervention (DOTSI).

SUMMARY:
This study evaluates the improvement of participation in everyday occupation among preschool children with mild developmental disabilities as a result of Occupational Therapy intervention.

DETAILED DESCRIPTION:
Preschoolers suffering from mild developmental disabilities are being referred to Occupational Therapy (OT) clinics according to limitation in participating of daily occupations. As well these children often demonstrate behavior or emotional difficulties. The primary treatment goal is promoting participation yet many times the treatment focuses on child's performance skills and not on occupation based activities. Respectively its outcome measures are the child performance skills. This study will document the therapeutic intervention, and evaluate its impact on child participation as well on his performance skills and emotional aspects. Participants will be recruited from waiting list for Occupational Therapy at Clalit Health services, Child Development Institute, and will be evaluate four times. First time on referral to waiting list ( At the present time due to long waiting list, children are waiting about three to four months before starting OT intervention), second time before treatment, third time after three of treatments and last follow-up after three months.

ELIGIBILITY:
Inclusion Criteria:

* kindergarten students of regular education
* Hebrew speaking

Exclusion Criteria:

* Students of special education
* Attending physiotherapy or psychology treatments
* Autistic Spectrum Disorder
* Cerebral Palsy
* Spina Bifida
* Developmental Intellectual Disabilities
* Blindness
* Deafness

Ages: 54 Months to 83 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Kindergarten's children referred to Occuptaion Therapy
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Improvement of child participation | up to 12 weeks
  Improvement of Participation of daily occupation as measured with Child Participation Questionnaire (CPQ)

SECONDARY OUTCOMES:
Child performance skills | up to 12 weeks
  Child Performance Skills Questionnaire (PSQ)
Child emotional aspects - Self efficacy | up to 12 weeks
  Pictorial scale of Perceived Competence and Social Acceptances for Young Children (PSPCSA)
Parental aspects- Parental self efficacy | up to 12 weeks
  Parental Efficacy Questionnaire
Child emotional aspects - Anxiety | up to 12 weeks
  Preschool Anxiety Scale (PAS)
Child emotional aspects - Mastery motivation | up to 12 weeks
  Dimension of Mastery Questionnaire (DMQ18)
Child performance skills -Fine motor precision | up to 12 weeks
  Bruininks-Oseretsky Test of Motor Proficiency (BOT2)
Child performance skills - Balance | up to 12 weeks
  Bruininks-Oseretsky Test of Motor Proficiency (BOT2)
Child performance skills -Executive functions | up to 12 weeks
  Day - Night task
Child performance skills - Sensory profile | up to 12 weeks
  Short Sensory Profile (SSP2)
Child performance skills -Core strength | up to 12 weeks
  Prone Extension Posture
Child performance skills - Visual motor integration | up to 12 weeks
  Developmental Test of Visual-Motor Integration (VMI)
Child performance skills - Draw a picture | up to 12 weeks
  Goodenough-Harris Drawing Test (DAP)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard G Robinson, Md, Principal Investigator — Clalit Health Services
Locations (1):
- Clalit Health Services, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No